CLINICAL TRIAL: NCT05176301
Title: Comparison Between the Coronal Diameters of the Cervical Spinal Canal and Spinal Cord Measured Using Computed Tomography and Magnetic Resonance Imaging in Korean Patients
Brief Title: Cervical Cord to Canal Diameter Ratio
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Jin Yong Jung, Professor, Daegu Catholic University Medical Center
Other Study IDs: DaeguCUMC
Record Dates: First submitted 2021-12-03; First posted 2022-01-04 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cervical Pain
Keywords: Coronal; Cervical canal diameter; Cervical cord diameter
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: computed tomography, Magnetic resonance image — Investigators measured the cervical cord and canal diameter by using CT and MRI that were previously taken.

SUMMARY:
Cervical epidural block could cause spinal cord injury if the epidural needle is over-inserted and punctures the spinal cord. Investigators retrospectively evaluated the imaging data of 100 patients (50 men and 50 women) who underwent both cervical computed tomography (CT) and cervical magnetic resonance imaging (MRI) at our hospital. Investigators measured the diameters of the spinal canal and spinal cord from the 3rd cervical vertebra to the 1st thoracic vertebra (T1) at each level by using the patients' cervical CT and MR images. The spinal cord and spinal canal diameters were measured in the transverse plane of cervical MR and CT images, respectively.

DETAILED DESCRIPTION:
The spinal canal diameter, i.e., the epidural transverse diameter, was measured as the distance between the innermost border of the left and right pedicles at each upper pedicular level from C3 to T1 on transverse CT images by using a picture archiving and communication system (PACS; INFINITT PACS G3, INFINITT Healthcare, Korea) The spinal cord diameter was measured between the left and right outermost distances of the cord at each upper pedicular level, which were almost the same locations used for measuring the spinal canal diameter, from C3 to T1 on transverse MR images by using the PACS.

ELIGIBILITY:
Inclusion Criteria:

* 100 patients (50 men and 50 women aged 20 to 70 years old) who visited our hospital and underwent both cervical CT and MRI simultaneously

Exclusion Criteria:

* patients who had a history of cervical spine surgery or cervical cord edema, whose CT or MR images did not include all the cervical vertebrae from C3 to T1,
* patients who had at least one missing medical detail such as diagnosis, age, height, or weight.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who visited Daegu catholic university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
the cord to canal diameter ratio | from December 1, 2020 through study completion, an average of 2 years were investigated retrospectively.
  the measurement of the cord to canal diameter ratio, i.e., the cord to epidural space diameter ratio of each cervical vertebral level from the 3rd cervical vertebra (C3) to the 1st thoracic vertebra (T1) in the coronal plane

CONTACTS AND LOCATIONS:
Overall Officials: Jin Y Jung, M.D., Study Chair — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No